CLINICAL TRIAL: NCT02350322
Title: Diet and Learning Abilities in Norwegian Youths
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Nutrition and Seafood Research, Norway (Other Government)
Collaborators: NORCE Norwegian Research Centre AS (Other); University of Tromso (Other)
Responsible Party: Principal Investigator, Lisbeth Dahl, PhD, National Institute of Nutrition and Seafood Research, Norway
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: FHF 900842 WP6
Record Dates: First submitted 2015-01-19; First posted 2015-01-29 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Cognitive Performance; Health Behavior; Nutrient Status
Keywords: Diet; concentration; seafood; youths; Norway; Nutrient status in blood; Inflammatory markers
MeSH Terms: conditions — Health Behavior | interventions — In Situ Hybridization, Fluorescence; Dietary Supplements

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Schoolmeal with fatty fish (Experimental): Fatty fish diet
  Interventions: Other: Schoolmeal with fatty fish
- Schoolmeal without fish (Experimental): Meat/cheese diet (non-seafood)
  Interventions: Other: Schoolmeal without fish
- Supplement (Experimental): Omega-3 capsules
  Interventions: Dietary Supplement: Supplement

INTERVENTIONS:
Other: Schoolmeal with fatty fish — Schoolmeal with fatty fish three times a week for 12 weeks
  Arms: Schoolmeal with fatty fish
Other: Schoolmeal without fish — Schoolmeal with meat/cheese three times a week for 12 weeks
  Arms: Schoolmeal without fish
Dietary Supplement: Supplement — Omega-3 capsules three times a week for 12 weeks
  Arms: Supplement

SUMMARY:
The aim of this study is to assess the effects of giving a schoolmeal with fatty fish, a schoolmeal without fish or omega-3 capsules on Noregian adolescents cognitive performance (concentration and learning abilities), mental health statua and markers of nutritional status. In addition, to disentangle the effect of fatty fish eaten as food and the effects of omega-3 fatty acids taken as a supplement.

DETAILED DESCRIPTION:
There has been an increased attention to the role of nutrition for learning abilities among schoolchildren. As the diet provides humans with energy and several essential nutrients, a balanced supply of all nutrients promotes not only physical growth and health, but also cognitive development, helping children to learn from infancy throughout adolescence and beyond. In a three-armed non-blinded intervention trial the investigators will test whether ingestion of a schoolmeal or omega-3 capsules will improve cognitive function among pupils in 9th grade at eight lower secondary school. The pupils will be randomised into three groups, one group will be served lunch with fatty fish, one group will be served similar lunch with meat/cheese (without fish) and one group will recieve omega-3 capsules three times week over a period of 12 weeks. At the beginning and at the end of the study, pupils should conduct cognitive tests, and blood-, urine- and hair samples will be taken. The pupils should also answer a questionnaire on their diet, physical activity, sleep pattern and mental health.

ELIGIBILITY:
Inclusion Criteria:

* girls and boys at lower secondary schools (9th grade)

Exclusion Criteria:

* allergy or intolerance to the food or food ingredients in the study

Ages: 14 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 478 (Actual)
Dates: Start 2015-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Concentration performance and literary skills | 12 weeks
  Age stanardardized d2 test of attention. Abilities in reading and spelleing through a Norwegain based intrument developed to evaluate the childrens literacy skills in the Norwegain language.

SECONDARY OUTCOMES:
Fatty acids | 12 weeks
  Levels of fatty acids in red blood cells before and after the intervention
Vitamin D status | 12 weeks
  Levels of 25-hydroxy vitamin D in serum blood before and after the intervention
Mental health | 12 weeks
  Mental health status measured by the Strengths and difficulties questionnaire (SDQ)
Iodine | 12 weeks
  Levels of iodine in urine samples before and after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Ingvild Eide Graff, PhD, Study Director — NIFES, PO Box 2029 Nordnes, N-5817 Bergen, Norway
Locations (1):
- Lisbeth Dahl, Bergen, Norway

REFERENCES:
- [Derived] Handeland K, Skotheim S, Baste V, Graff IE, Froyland L, Lie O, Kjellevold M, Markhus MW, Stormark KM, Oyen J, Dahl L. The effects of fatty fish intake on adolescents' nutritional status and associations with attention performance: results from the FINS-TEENS randomized controlled trial. Nutr J. 2018 Feb 23;17(1):30. doi: 10.1186/s12937-018-0328-z. PMID 29475446
- [Derived] Handeland K, Oyen J, Skotheim S, Graff IE, Baste V, Kjellevold M, Froyland L, Lie O, Dahl L, Stormark KM. Fatty fish intake and attention performance in 14-15 year old adolescents: FINS-TEENS - a randomized controlled trial. Nutr J. 2017 Oct 2;16(1):64. doi: 10.1186/s12937-017-0287-9. PMID 28969711